CLINICAL TRIAL: NCT02018705
Title: Comparison of Peroral Endoscopic Myotomy (POEM) With Laparoscopic Heller Myotomy (LHM) for Treatment of Achalasia, a Retrospective Multicenter Study
Brief Title: Comparison of Peroral Endoscopic Myotomy (POEM) With Laparoscopic Heller Myotomy (LHM) for Treatment of Achalasia
Acronym: POEM3
Status: Terminated | Type: Observational
Why Stopped: data income too low
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Agaplesion Markus Krankenhaus (Unknown); Johannes Gutenberg University Mainz (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); McGill Faculty of Medicine (Unknown); University Hospital, Zürich (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Medical Director, Interdisciplinary Endoscopy Department and Clinic, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV4519; Ethics Committee, Hamburg (Registry Identifier: PV 4519)
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Comparison of Short- Term Success Rates of POEM With LHM; Comparison of Long-term Success Rates of POEM With LHM
Keywords: POEM; LHM; Achalasia treatment; LES sphincter myotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- POEM: group of Achalasia patients treated with POEM (peroral endoscopic myotomy)
- LHM: group of Achalasia patients treated with LHM (laparoscopic Heller myotomy)(+ fundoplication)

SUMMARY:
For the treatment of Achalasia, LHM has been the only surgical therapy. Recently, an endoscopic approach for this therapy has been developed (peroral endoscopic Myotomy POEM). Studies show promising short and mid term results for POEM. At present, POEM is considered a promising new technique with the potential to become a standard achalasia treatment. For this to happen, long-term comparative data with LHM is required. Therefore,the intention for this study is to investigate the short and long-term efficacy of POEM for the treatment of achalasia as it was performed in international centers and compare outcomes with database assessment of LHM.

DETAILED DESCRIPTION:
Achalasia is a neurodegenerative esophageal motility disorder characterized by incomplete lower esophageal sphincter (LES) relaxation, increased LES tone, and aperistalsis of the esophagus. The standard surgical treatment for achalasia is laparoscopic Heller Myotomy (LHM). A recent meta-analysis of 105 studies reporting on 7855 patients demonstrated that laparoscopic Heller myotomy is the most effective and long-lasting therapy for achalasia. Superior to Endoscopic balloon dilatation or Botulinumtoxin injection LHM has a one year therapeutic efficacy in approximately 90% of patients. Recently an endoscopic technique emulating the principles of LHM was developed. This technique of a purely endoscopic myotomy has been demonstrated by Pasricha et al. in animal experiments and Inoue et al. reported the first clinical study. Other pilot studies and a larger international multi-center trial have replicated promising results for POEM.

Uncontrolled studies show promising short and mid term results for POEM. At present, POEM is considered a promising new technique with the potential to become a standard achalasia treatment. For this to happen, however, comparative data with LHM is required. Our study group intends to investigate the short and long-term efficacy of POEM for the treatment of achalasia as it was performed in international centers and compare outcomes with database assessment of LHM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic achalasia and pre-op barium swallow, manometry and oesophago-gastro-duodenoscopy which have been consistent with the diagnosis
* Age > 18 years with medical indication for interventional achalasia treatment
* Availability of Eckardt score at baseline and 12 months after initial treatment

Exclusion Criteria:

* Patients with previous surgery of the stomach or esophagus
* Patients with known coagulopathy
* Previous surgical achalasia treatment
* Patients with liver cirrhosis and/or esophageal varices
* Active esophagitis
* Eosinophilic esophagitis
* Barrett's esophagus
* Stricture of the esophagus
* Malignant or premalignant esophageal lesion
* Severe Candida esophagitis
* Hiatal hernia > 1cm
* Extensive, tortuous dilatation (>7cm luminal diameter, S shape) of the esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Achalasia patients who have been treated with either POEM or LHM
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
treatment success | 1 year after treatment
  treatment success is defined as an Eckardt Score </=3

SECONDARY OUTCOMES:
procedure related adverse events | 3 months after treatment
  retrospective data for this timepoint can be used of the interval 2-8 months after the initial procedure
lower esophageal sphincter pressure (LESP) | 3 months after treatment
  retrospective data for this timepoint can be used of the interval 2-8 months after the initial procedure
symptomatic reflux and use of antacid medication | 3 months after treatment
  retrospective data for this timepoint can be used of the interval 2-8 months after the initial procedure
procedure related adverse events | 12 months after treatment
  retrospective data for this timepoint can be used of the interval 9-15 months after the initial procedure
lower esophageal sphincter pressure (LESP) | 12 months after treatment
  retrospective data for this timepoint can be used of the interval 9-15 months after the initial procedure
symptomatic reflux and use of antacid medication | 12 months after treatment
  retrospective data for this timepoint can be used of the interval 9-15 months after the initial procedure

OTHER OUTCOMES:
any reported GERD data | procedure to five years after treatment
duration of procedure | procedure
  duration of procedure (minutes)
in-hospital stay | procedure
  in-hospital stay of patients (days)
length of myotomy | procedure
  length of myotomy (centimeters)
procedure related complications | procedure
  any complication during performance of treatment that required conversion to either laparoscopic (POEM) or open surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — University Hospital Eppendorf, Hamburg
Locations (5):
- Aarhus University Hospital, Aarhus, Denmark
- Germany (2):
  - University Hospital Eppendorf, Hamburg
  - University Medical Center, Mainz
- Academic Medical Center, Amsterdam, Netherlands
- University Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Campos GM, Vittinghoff E, Rabl C, Takata M, Gadenstatter M, Lin F, Ciovica R. Endoscopic and surgical treatments for achalasia: a systematic review and meta-analysis. Ann Surg. 2009 Jan;249(1):45-57. doi: 10.1097/SLA.0b013e31818e43ab. PMID 19106675
- [Background] Pasricha PJ, Hawari R, Ahmed I, Chen J, Cotton PB, Hawes RH, Kalloo AN, Kantsevoy SV, Gostout CJ. Submucosal endoscopic esophageal myotomy: a novel experimental approach for the treatment of achalasia. Endoscopy. 2007 Sep;39(9):761-4. doi: 10.1055/s-2007-966764. PMID 17703382
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] Zhou PH, Li QL, Yao LQ, Xu MD, Chen WF, Cai MY, Hu JW, Li L, Zhang YQ, Zhong YS, Ma LL, Qin WZ, Cui Z. Peroral endoscopic remyotomy for failed Heller myotomy: a prospective single-center study. Endoscopy. 2013;45(3):161-6. doi: 10.1055/s-0032-1326203. Epub 2013 Feb 6. PMID 23389963
- [Background] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665
- [Background] Von Renteln D, Fuchs KH, Fockens P, Bauerfeind P, Vassiliou MC, Werner YB, Fried G, Breithaupt W, Heinrich H, Bredenoord AJ, Kersten JF, Verlaan T, Trevisonno M, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: an international prospective multicenter study. Gastroenterology. 2013 Aug;145(2):309-11.e1-3. doi: 10.1053/j.gastro.2013.04.057. Epub 2013 May 9. PMID 23665071
- [Background] Swanstrom LL, Rieder E, Dunst CM. A stepwise approach and early clinical experience in peroral endoscopic myotomy for the treatment of achalasia and esophageal motility disorders. J Am Coll Surg. 2011 Dec;213(6):751-6. doi: 10.1016/j.jamcollsurg.2011.09.001. Epub 2011 Oct 13. PMID 21996484
- [Background] Costamagna G, Marchese M, Familiari P, Tringali A, Inoue H, Perri V. Peroral endoscopic myotomy (POEM) for oesophageal achalasia: preliminary results in humans. Dig Liver Dis. 2012 Oct;44(10):827-32. doi: 10.1016/j.dld.2012.04.003. Epub 2012 May 19. PMID 22609465